CLINICAL TRIAL: NCT05158972
Title: Observational Study to Evaluate the Actual Use and Effectiveness of Dymista® Nasal Spray in Asian Patients
Status: Completed | Type: Observational
Sponsor: Mylan Inc. (Industry)
Collaborators: MEDA Pharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Other Study IDs: 3325
Record Dates: First submitted 2021-10-26; First posted 2021-12-15 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-05

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dymista®: Dymista® (Azelastine hydrochloride and Fluticasone propionate) nasal spray as prescribed within routine clinical practice
  Interventions: Drug: Dymista

INTERVENTIONS:
Drug: Dymista — 1 spray per nostril twice daily up to four weeks

SUMMARY:
Gathering knowledge on the use of Dymista® in Asian patients who receive Dymista® for the first time in routine clinical practice

DETAILED DESCRIPTION:
A) Primary objective:

Gathering knowledge on the use of Dymista® in Asian patients who receive Dymista® for the first time in routine clinical practice; Patient's demographic;

Anamnestic background including:

* allergic and other comorbidities
* allergic conjunctivitis
* polysensitization
* current symptoms
* previous treatments of allergic rhinitis
* usage of current asthma reliever medication
* family history of allergy

B) Secondary Objective:

* Response to therapy with Dymista® nasal spray in routine clinical practice.
* Quality of sleep (by VAS)
* Troublesomeness in daily activities (by VAS)
* Patient's assessment about the regular use of Dymista®
* Patients opinion about continuation of Dymista® treatment after end of the observational period

ELIGIBILITY:
Inclusion Criteria:

* The first prescription of Dymista® nasal spray according to the summary of product characteristics (SPC) and patient information leaflet and independently from the patient's enrollment in the study.
* Patients with moderate to severe seasonal or perennial allergic rhinitis
* For Hong Kong and Malaysia: Adult and children of age ≥ 12 years
* For Taiwan: Adult and children of age ≥ 6 years.
* For Thailand: Adults and children of age ≥ 12 years with seasonal and/or perennial allergic rhinitis OR children of age 6-11 years with only seasonal allergic rhinitis
* Acute allergic rhinitis symptoms at the day of inclusion (i.e. VAS-Score ≥50 mm)
* Signed informed consent/assent from the patient and, if applicable, the parent(s) or legal guardian(s) in compliance with local requirements.
* Ability to understand and follow the instructions for using Dymista® nasal spray according to the patient information leaflet.
* Willingness to complete and return the Patient Card.

Exclusion Criteria:

* VAS score <50 mm on day of inclusion
* Known allergic reaction from and/or intolerance to Dymista® nasal spray or any of the ingredients.
* Pregnancy/planned pregnancy or breastfeeding during this NIS
* Patients or parent(s)/legal guardians (as applicable) not able to fulfill study requirements according to the Investigator's opinion.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Use of Dymista® in Asian patients (Taiwan, Malaysia, Hongkong and Thailand) with moderate to severe seasonal or perennial allergic rhinitis under real life conditions.
Sampling Method: Non-Probability Sample
Enrollment: 924 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Profile of Asian AR patients prescribed with Dymista® | The duration of the study is approximately 28 days after the eligible patients or caregivers provided the written informed consent
  The primary outcome of this non-interventional study is the exploratory description of patient characteristics in regard to demographics, symptoms and allergic rhinitis phenotypes in real life receiving Dymista for the first time.

SECONDARY OUTCOMES:
Effectiveness of Dymista® in Asian AR patients (Symptom Severity Assessment by VAS) | From day 1 to day 28
  Response to treatment would be assessed by self-reported severity of symptoms (change of Visual Analog Score). The visual analog scale titled as "Please reflect how much bothersome your OVERALL allergic rhinitis symptoms were within the previous 24 hours" This will be done by marking with a pen the printed visual analog scale over the patient card at the appropriate range (not at all bothersome / troubled = 0 to extremely bothersome / troubled = 100 mm).
Effectiveness of Dymista® in Asian AR patients (QOL assessment by VAS) | From day 1 to day 28
  Sleep change will be assessed by self-reported quality of sleep (change of Visual Analog Score). The visual analog scale titled as "Please reflect how troubled you have been by lack of good night sleep during the previous 7 days as a result of your allergic rhinitis symptoms." This will be done by marking with a pen the printed visual analog scale over the patient card at the appropriate range (not at all bothersome / troubled = 0 to extremely bothersome / troubled = 100 mm).
Effectiveness of Dymista® in Asian AR patients (Impact on daily activities assessment by VAS) | From day 1 to day 28
  Impact on daily activities will be assessed by self-reported troubles in daily activities (change of Visual Analog Score). The visual analog scale titled as "Please reflect how troubled you have been by the following activities (Regular activities at home and work / school, Social activities, Outdoor activities) during the previous 7 days as a result of your allergic rhinitis symptoms".
  For each of these activities, it will be done by marking with a pen the printed visual analog scale over the patient card at the appropriate range (not at all bothersome / troubled = 0 to extremely bothersome / troubled = 100 mm).

CONTACTS AND LOCATIONS:
Locations (33):
- Hong Kong (2):
  - Hong Kong ENT Clinic, Hong Kong
  - Asia Priority Healthcare, Kowloon
- Malaysia (8):
  - Kempas Medical Center, Johor Bahru
  - KPJ Johor Specialist Hospital, Johor Bahru
  - Allergy and Immunology Clinic Gleneagles Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Universiti Sains Malaysia, Kubang Kerian
  - Sarawak General Hospital, Kuching
  - Pantai Hospital Ipoh, Perai
  - Hospital Sultan Abdul Aziz Shah, Serdang
- Taiwan (9):
  - St. Martin De Porres Hospital, Chiayi City
  - Chang Gung Memorial Hospital-KAOHSIUNG, Kaohsiung City
  - Asia University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Municipal Wan Fang Hospital, Taipei
  - China Medical University Hsinchu Hospital, Zhubei
- Thailand (14):
  - Bangkok hospital, Bangkok
  - King Chulalongkorn Memorial Hospital (Department of Medicine), Bangkok
  - King Chulalongkorn Memorial Hospital (Department of Pediatrics), Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Ramathibodi hospital, Bangkok
  - Siriraj Hospital (Department of Medicine), Bangkok
  - Siriraj Hospital (Department of Otorhinolaryngology), Bangkok
  - Thammasat University Hospital (Department of Otolaryngology), Bangkok
  - Thammasat University Hospital (Department of Pediatrics), Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Naresuan University Hospital, Phitsanulok
  - Songkla University Hospital, Songkhla

IPD SHARING:
Plan to Share IPD: No